CLINICAL TRIAL: NCT03264261
Title: Constraint Induced Movement Therapy for Walking in Individuals Post Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Ming Wu, Research Scientist, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD082216 (NIH)
Record Dates: First submitted 2017-08-14; First posted 2017-08-29 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Stroke
Keywords: stroke, locomotion
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Subjects will be blocked by gait speed into slow (< 0.4 m/s) or fast (≥ 0.4 m/s) subgroups and randomized to either the CIMT or treadmill training only groups at the initial test.
Who Masked: Outcomes Assessor
Masking Description: Outcome measures of each subject will be evaluated before training, after 6 weeks of training, and at 8 weeks after the end of training by a physical therapist who is blinded by subject group assignment, and subjects will be requested not to disclose his/her group assignment to this physical therapist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- robotic training (Experimental): For the robotic training group, a controlled resistance load will be applied to the unaffected leg at the ankle and an assistance load will be applied to the pelvis.
  Interventions: Device: robotic training
- treadmill training (Active Comparator): For the treadmill training only group, a physical therapist will provide manual assistance to the affected leg at the knee and/or ankle joints as necessary during treadmill training.
  Interventions: Device: treadmill training

INTERVENTIONS:
Device: robotic training — robotic training, 3 times/week for 6 weeks
  Arms: robotic training
Device: treadmill training — treadmill training only, 3 times/week for 6 weeks
  Arms: treadmill training

SUMMARY:
To compare the effect of constraint induced movement therapy (CIMT) vs. treadmill training only on walking function in individuals post-stroke, a 6 week, single-blind, randomized training study will be conducted with three assessments of gait to determine the training effect. Subjects will be randomized to either the CIMT or treadmill training only groups at the initial test. Following the initial test, individuals from the 2 groups will undergo intensive locomotor training. Training will be performed 3 times per week for 6 weeks with the training time for each visit set to 45 minutes as tolerated. Data collection will proceed until 36 subjects from 2 groups have been trained.

DETAILED DESCRIPTION:
To determine the effect of constraint induced movement therapy (CIMT) on locomotor function in individuals post stroke. In order to compare the effect of CIMT vs. treadmill training only on walking function in individuals post-stroke, a 6 week, single-blind, randomized training study will be conducted with three assessments of gait to determine the training effect. Subjects will be blocked by gait speed into slow (< 0.4 m/s) or fast (≥ 0.4 m/s) subgroups and randomized to either the CIMT or treadmill training only groups at the initial test. Following the initial test, individuals from the 2 groups will undergo intensive locomotor training. Training will be performed 3 times per week for 6 weeks with the training time for each visit set to 45 minutes as tolerated, excluding set up time. Data collection will proceed until 36 subjects from 2 groups have been trained.

ELIGIBILITY:
Inclusion Criteria:

1. age between 21 and 75 years;
2. history of unilateral, supratentorial, ischemic or hemorrhagic stroke;
3. no prior stroke;
4. demonstration of impaired walking function (self-selected walking speed ≤ 0.80 m/s);
5. able to stand and walk (>10 meters) without physical assistance.

Exclusion Criteria:

1. significant cardiorespiratory/metabolic disease;
2. other neurological or orthopedic injury that impairs locomotion;
3. scores on the Mini Mental Status examination < 24;
4. stroke of the brainstem or cerebellar lesions;
5. uncontrolled hypertension (systolic > 200 mm Hg, diastolic > 110 mm Hg);
6. botox injection within 6 months of starting the study.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-08-14 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in walking speed | pre, post 6 weeks training, and 8 weeks after the end of training.
  Overground gait speed will be collected on a 10 m instrumented walkway
Change in 6-minute walking distance | pre, post 6 weeks training, and 8 weeks after the end of training.
  walking distance covered by subjects in 6 minutes

SECONDARY OUTCOMES:
Change in Berg Balance Scale | pre, post 6 weeks training, and 8 weeks after the end of training.
  Berg Balance Scale scores will be collected by research physical therapist

CONTACTS AND LOCATIONS:
Overall Officials: Ming Wu, PhD, Principal Investigator — Abilitylab
Locations (1):
- Abilitylab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No